CLINICAL TRIAL: NCT04354675
Title: A Randomized Trial Comparing the Effectiveness of Pre-test Genetic Counseling Using an Artificial Intelligence Program and Traditional In-person Genetic Counseling in Women Newly Diagnosed With Breast Cancer Who do Not Currently Meet National Comprehensive Cancer Network (NCCN) Criteria for Genetic Testing.
Brief Title: Effectiveness of AI Genetic Counseling Program vs In-person Genetic Counseling in Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CASE12119
Record Dates: First submitted 2020-03-25; First posted 2020-04-21 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial intelligence program (Experimental): Will complete consult with the use of an artificial intelligence program Chatbot.
  Interventions: Genetic: Automated program (ChatBot); Other: BCGCKQ Survey; Other: Satisfaction Survey; Device: Genetic testing
- in-person genetic counseling (Active Comparator): Will complete a traditional in-person genetic counseling. consult by meeting with a Genetics Counselor
  Interventions: Genetic: Genetics counselor; Other: BCGCKQ Survey; Other: Satisfaction Survey; Device: Genetic testing

INTERVENTIONS:
Genetic: Automated program (ChatBot) — Pre-test counseling and information through a pre-test automated genetic counseling program (ChatBot)
  Arms: Artificial intelligence program
Genetic: Genetics counselor — Traditional in-person genetic counseling
  Arms: in-person genetic counseling
Other: BCGCKQ Survey — Survey assessing Breast Cancer Genetic Counseling Knowledge Questionnaire (BCGCKQ)
  Other Names: Breast Cancer Genetic Counseling Knowledge Questionnaire (BCGCKQ)
Other: Satisfaction Survey — Survey assessing satisfaction with Decision-Genetic Testing
Device: Genetic testing — Genetic testing for all participants will assess for a mutation in 47 genes commonly associated with hereditary cancer syndromes (Invitae's Common Hereditary Cancer Panel) for those who choose to complete testing.

SUMMARY:
The purpose of this study is to help better understand the uptake and impact of genetic testing for women diagnosed with breast cancer who do not meet National Comprehensive Cancer Network (NCCN) criteria for genetic testing. By doing so, the research team will gain a better understanding of the clinical implications for offering genetic testing for all patients recently diagnosed with breast cancer versus only offering genetic testing to those meeting NCCN criteria.

By offering genetic counseling and genetic testing to all women recently diagnosed with breast cancer, there will be a shortage of genetic counselors. This study will also assess the feasibility of using artificial intelligence to assist in the genetic counseling process.

DETAILED DESCRIPTION:
This is a randomized trial comparing the effectiveness of pre-test genetic counseling using an artificial intelligence program and traditional in-person genetic counseling in women newly diagnosed with breast cancer who do not currently meet National Comprehensive Cancer Network (NCCN) criteria for genetic testing.

The primary objectives of this study are:

1. To determine up-take of testing for those who do not meet NCCN guidelines for genetic testing
2. To assess overall patient satisfaction and comprehension in both groups

The secondary objectives of this study are:

1. To assess mutation rate in the overall cohort
2. Identify reasons for not pursuing genetic testing
3. Identify any specific areas of improvement in satisfaction and comprehension
4. Assess the impact of genetic testing on Time to Treatment in this cohort
5. Develop workflow for offering genetic testing, providing pre-test genetic counseling, ordering testing, and delivering results

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with Stage 0-3 breast cancer.
* Patients who do not satisfy current NCCN criteria for referral to a genetics counselor and genetics testing.
* Must have the ability to understand and the willingness to sign a written informed consent document as well as complete the study questionnaires.

Exclusion Criteria:

- N/A

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent of participants who took up genetic testing after not meeting NCCN guidelines for genetic testing | 2 years
  Up-take of testing for those who do not meet NCCN guidelines for genetic testing
Mean overall patient satisfaction with decision about genetic testing: survey | 2 years
  Mean overall patient satisfaction with decision about genetic testing as assessed by survey. The survey is a previously validated six-question Likert scale based survey. The scale ranges from 6 to 30, with higher scores indicating more satisfaction.
  Satisfaction will be compared between groups with t-test or Wilcoxon rank sum test. Published data suggest that standard deviation on the satisfaction survey is 3. A 2 point difference in average satisfaction score between groups is considered to be relevant
Overall comprehension as assessed by BCGCKQ | 3 years
  Comprehension as assessed by previously validated survey consisting of 27 questions, which are a blend of True or False and multiple choice questions. The scale ranges from to , with higher scores indicating more comprehension.
  Comprehension will be compared between groups with t-test or Wilcoxon rank sum test.

SECONDARY OUTCOMES:
Percentage of overall cohort with mutation | 2 years
  Mutation rate as described by percentage of overall cohort with mutation. Groups will be compared with Chi-square test or Fisher's exact test
Number of patients who decline genetic testing | 2 years
  Number of patients who decline genetic testing. Groups will be compared with Chi-square test or Fisher's exact test
Frequencies of most common reasons for not pursuing genetic testing | 2 years
  Reasons for not pursuing genetic testing in those who declined will be collected as a descriptive measure and then analyzed as frequencies of the different responses, summarizing the most common answers
Time to treatment | 3 years
  Time to treatment will be compared between patients who had genetic testing to those who did not using t-test or Wilcoxon rank sum test among all study patients.

CONTACTS AND LOCATIONS:
Overall Officials: Zahraa Al-Hilli, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Commercially available software being used to conduct the study